CLINICAL TRIAL: NCT05935267
Title: Thoracostomy Tube Irrigation: a Multi-Center Trial Investigating Its Efficacy in the Reduction of Secondary Intervention for the Management of Retained Hemothorax
Brief Title: Thoracostomy Tube Irrigation: a Multi-Center Trial
Status: Active, not recruiting | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 039.GME.2021.D
Record Dates: First submitted 2022-02-21; First posted 2023-07-07 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Thoracic Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- control cohort: control cohort
  Interventions: Procedure: thoracic irrigation
- irrigation cohort: irrigation cohort
  Interventions: Procedure: thoracic irrigation
- standard cohort: standard cohort
  Interventions: Procedure: thoracic irrigation

INTERVENTIONS:
Procedure: thoracic irrigation — We will start this study using 20% as the approximate national intervention rate, based on current literature, with the goal of detecting a 50% reduction in the experimental arm (i.e. 10% secondary intervention rate after thoracic irrigation). Therefore, we will plan to enroll 108 patients in the irrigation cohort and 324 patients in the control cohort. An interim analysis will be conducted once 54 patients have been enrolled in the irrigation cohort. The secondary intervention rate in the irrigation cohort and the standard cohort will be determined, and any adjustments to sample size will be made at that time.

SUMMARY:
All trauma patients ages 18 years or older presenting within 24 hours of blunt or penetrating injury resulting in traumatic HTx or HPTx will be eligible for enrollment. This prospective comparative study will consist of a non-irrigation control arm and a thoracic irrigation experimental arm. Thoracic irrigation is performed at the time of the initial TT placement, and is done at the discretion of the attending Trauma surgeon. All patients enrolled will be entered in a prospectively maintained thoracic trauma database. The primary outcome is need for secondary intervention, defined as additional TT placement, VATS, tissue plasminogen activator (tPA), or thoracotomy for the management of retained HTx. Secondary interventions will be screened according to indication. Only secondary interventions directed at management of retained collection will be considered in the analysis for our primary outcome. Secondary intervention aimed at persistent air leaks or post-pull PTx will be considered separately in any analysis.

DETAILED DESCRIPTION:
All trauma patients ages 18 years or older presenting within 24 hours of blunt or penetrating injury resulting in traumatic HTx or HPTx will be eligible for enrollment. This prospective comparative study will consist of a non-irrigation control arm and a thoracic irrigation experimental arm. Thoracic irrigation is performed at the time of the initial TT placement, and is done at the discretion of the attending Trauma surgeon. All patients enrolled will be entered in a prospectively maintained thoracic trauma database. The primary outcome is need for secondary intervention, defined as additional TT placement, VATS(Viral Activation Transfusion Study), tissue plasminogen activator (tPA), or thoracotomy for the management of retained HTx. Secondary interventions will be screened according to indication. Only secondary interventions directed at management of retained collection will be considered in the analysis for our primary outcome. Secondary intervention aimed at persistent air leaks or post-pull PTx will be considered separately in any analysis.

This is a multicenter observational prospective data collection study. The study was initiated by Dr. Carver at the Medical College of Wisconsin and hosted as a Western Trauma Association Multicenter trial. We will not alter our standard of care practice at Methodist Dallas Medical Center in any way during the study duration. Data abstraction will occur from the electronic medical records program (EPIC). Each participating site will also practice according to their standard of care. If a site chooses to implement a TT irrigation protocol, approval should be obtained from their local divisional and IRB(Institutional Review Board) committees. If a participating site already performs thoracic irrigation, efforts should be made to follow the TT irrigation protocol provided with this study.

Each participating site will develop a method to screen for patients based on the resources available at their institution; this method should be included in the proposal submitted to their IRB.

The data at each participating site will be collected by a member of the study team and entered into the secure REDCap (Research Electronic Data Capture) database specifically created for this project. Data will be transferred from participating sites to Medical College of Wisconsin via REDCap. REDCap is a secure web application for building and managing online databases. All data entered into REDCap and transferred between sites will be deidentified. Only approved study staff at each site will be granted password protected access to the REDCap database. Ultimately, the Medical College of Wisconsin PI will have control over who can access the database and what type of access is granted.

The aim is to have all data collection completed by December 31, 2022 and to have data analysis completed by July 1, 2022.

ELIGIBILITY:
Inclusion Criteria:

* • Trauma patients admitted with initial indication for TT placement of HTx or HPTx.

  * Patients must present to Methodist Dallas Medical Center within 24 hours of the traumatic event, either blunt or penetrating injury.
  * Follow up data available including radiologic studies performed within 24 hours of tube placement and hospital records to determine if any additional intervention(s) was performed.
  * 18 years of age or older.

Exclusion Criteria:

* Less than 18 years of age.
* Patients who had the TT removed (intentionally or unintentionally dislodged) prior to 24 hours TT duration.
* Patients requiring operative exploration of the thoracic cavity within 6 hours following TT placement.
* Patients with thoracotomy or VATS as initial treatment for HTx and/or HPTx
* Patients with TT placed for isolated PTx
* Patients who have a TT placed for HTx or HPTx more than 24 hours after presentation, or more than 24 hours after their traumatic event
* Pregnant or lactating women
* Prisoners
* Physician discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All trauma patients ages 18 years or older presenting within 24 hours of blunt or penetrating injury resulting in traumatic HTx or HPTx will be eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-12-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with thoracic trauma | Dec 2022 - Dec 2023
  thoracic trauma resulting in the formation of pneumothorax (PTx), hemothorax (HTx), or hemopneumothorax (HPTx) is successfully managed with thoracostomy tube (TT) placement to evacuate blood and / or air from the pleural space.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Truitt, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Clinical Research Institute Methodist Health System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided